CLINICAL TRIAL: NCT02519504
Title: Intervention and Outcomes in Duarte Galactosemia
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Judith Fridovich-Keil, Professor, Emory University
Other Study IDs: IRB00081271
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Duarte Galactosemia
Keywords: Galactose-1-phosphate uridylyltransferase deficiency; Cognitive disorders
MeSH Terms: conditions — Galactosemias; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Duarte galactosemia: Pediatric subjects with Duarte galactosemia will undergo direct assessments of cognitive skills (memory, executive function, and auditory processing), communication processes (speech and language), physical development (including motor skills, coordination, and occurrence of tremors), and social-emotional development.
- Control: Pediatric subjects without Duarte galactosemia will undergo direct assessments of cognitive skills (memory, executive function, and auditory processing), communication processes (speech and language), physical development (including motor skills, coordination, and occurrence of tremors), and social-emotional development.

SUMMARY:
The purpose of this study is to learn about Duarte galactosemia (DG). This study will examine the possible effects of Duarte galactosemia (DG) in children, and determine whether dietary exposure to milk in infancy or early childhood is associated with developmental outcomes of school-age children with Duarte galactosemia (DG).

DETAILED DESCRIPTION:
Duarte galactosemia (DG) is an autosomal recessive genetic condition characterized by partial loss of galactose-1-phosphate uridylyltransferase (GALT), which results in partially impaired metabolism of the sugar, galactose, which is abundant in milk and also found at lower levels in many other foods. There is currently no consensus on long-term outcome prognosis for infants with Duarte galactosemia (DG) and some studies suggest these children might be at increased risk for developmental difficulties later in childhood. There is also no conclusive data on whether children with Duarte galactosemia (DG) might benefit from dietary restriction of galactose. The investigator will be assessing whether 6-12 year old children with Duarte galactosemia experience developmental disorders relative to controls, and if so, whether dietary exposure to milk in infancy or early childhood is associated with developmental outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Healthy Children/Children with Duarte Galactosemia:

* Age between 6-12 years

Exclusion Criteria:

* Chronic illness
* Any condition unrelated to Duarte Galactosemia but known to cause developmental problems
* Children who did not have the current parent/guardian as the primary caregiver when the child was an infant

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study participants will be recruited in multiple collaborating states from records of infants born in that state who were diagnosed with Duarte Galactosemia detected by newborn screening (NBS). The current list of collaborating states includes: AL, CA, GA, IA, IL, MI, MO, NC, NJ, OR, SC, TX, WA, and WI but this list may change.
Sampling Method: Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Fridovich-Keil, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were recruited through collaboration with state new born screening programs or metabolic clinics. Those expressing interest were evaluated for eligibility and asked to complete an online survey.
Pre-assignment Details: Interest in participating was expressed by parents or caregivers for 600 children. Consent to participate was not given for 22 and consent was given for another 12 but the initial online survey was not completed.The case/control status and demographic information is unknown for these 34 children.
Groups:
- Children With Duarte Galactosemia (Cases): Pediatric subjects with Duarte galactosemia undergoing direct assessments of cognitive skills (memory, executive function, and auditory processing), communication processes (speech and language), physical development (including motor skills, coordination, and occurrence of tremors), and social-emotional development.
- Unaffected Siblings (Controls): Pediatric subjects without Duarte galactosemia undergoing direct assessments of cognitive skills (memory, executive function, and auditory processing), communication processes (speech and language), physical development (including motor skills, coordination, and occurrence of tremors), and social-emotional development.
Period: Overall Study
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Started (Completed the initial online survey) | 319 | 247
Attended Direct Testing | 212 | 149
Completed (Had complete information from the direct testing visit.) | 206 | 144
Not Completed | 113 | 103
Not completed — Protocol Violation | 6 | 5
Not completed — Ineligible for direct testing | 12 | 12
Not completed — Did not participate in direct testing | 95 | 86

BASELINE CHARACTERISTICS:
Population: Children completing the study are included in the baseline analysis population descripton.
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls) | Total
Number analyzed (Participants) | 206 | 144 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 206 | 144 | 350
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.39 (1.98) | 9.30 (1.84) | 9.36 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 65 | 158
  Male | 113 | 79 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 202 | 137 | 339
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 192 | 134 | 326
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 206 | 144 | 350
Breastmilk exposure [Count of Participants; unit: Participants]
  No breastmilk | 66 | 35 | 101
  Minimal breastmilk | 75 | 17 | 92
  Moderate breastmilk | 26 | 33 | 59
  Exclusively fed breastmilk | 39 | 59 | 98

OUTCOME MEASURES:

1. Primary Outcome: Children's Memory Scale Score
Description: The Children's Memory Scale assesses memory and learning across three domains: auditory/verbal, visual/nonverbal, and attention/concentration. Each domain contains two core subtests and one supplemental subtest, each of which contain both an immediate and delayed memory portion. From these subtests, eight Index scores are derived: Visual Immediate, Visual Delayed, Verbal Delayed, Verbal Delayed, Delayed Recognition, Overall Learning, Attention/Concentration, and General Memory. The Index scores represent functioning within and across the domains. The scaled scores of the subtests relevant to each Index score are summed, and from this sum, a normed Index score is derived. Each Index score has a range of 50-150, and an average score of 100, with most children scoring between 85 and 115 (SD=15). Lower scores indicate impaired memory abilities.
Time Frame: Baseline
Population: There were 2 occasions where due to unforeseen scheduling issues the study team was not able to do the psych testing on 2 control participants, this applies to all outcome measures with 142 controls instead of 144.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
score on a scale
  Visual Immediate Subtest | 106.76 (13.18) | 104.15 (12.88)
  Visual Delayed Subtest | 105.99 (12.19) | 103.78 (13.54)
  Verbal Immediate Subtest | 103.23 (16.20) | 103.08 (15.34)
  Verbal Delayed Subtest | 103.30 (15.53) | 104.35 (15.66)
  General Memory Index | 107.88 (14.05) | 106.40 (15.49)
  Attention/Concentration Subtest | 102.15 (15.32) | 104.86 (16.51)
  Learning Subtest | 104.16 (13.59) | 102.87 (14.65)
  Delayed Recognition Subtest | 102.88 (13.55) | 103.10 (15.08)

2. Primary Outcome: Wechsler Intelligence Scale for Children IV-Integrated (WISC-IV-Integrated): Digit Span Score
Description: Auditory working memory can be assessed using WISC-IV-Integrated: Digit Span test. The digit span test forward assesses attention and short-term memory while the digit span test backward assesses working memory. For the forward test, the examinee listens while examiner says a series of numbers and asks the participant to repeat them back in the same order. For the backward test, the examiner will ask the examinee to repeat the numbers backwards, that is, by starting with the last number said and going backwards to the first number said. This process continues until the examinee can no longer remember either the full sequence of numbers or the correct order. Both forward and reverse trials are given twice. The Digit Span test is scored by the amount of numbers the examinee was able to remember in each test. Scores could range from 0 to 16 with higher scores indicating better performance.
Time Frame: Baseline
Population: This assessment was not administered during the study because it was redundant to other tests already being used.
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Wechsler Intelligence Scale for Children IV-Integrated (WISC-IV-Integrated): Spatial Span Score
Description: Spatial working memory was assessed using the Wechsler Intelligence Scale for Children IV-Integrated (WISC-IV-Integrated): Spatial Span During the forward task, participants are presented with a board containing blue blocks randomly arranged. The rater first taps out a pattern of blocks, beginning with two blocks and increasing the number of blocks in the pattern with participant proficiency, and the participant is tasked with tapping the same pattern. For the backwards test, the participant is tasked with tapping out the reverse pattern after the rater's demonstration. These patterns also begin with two blocks and increase with participant proficiency. The score is the number of patterns completed correctly. Scores can range from 0 to 16 with higher scores indicating better performance.
Time Frame: Baseline
Population: There were 2 occasions where, due to unforeseen scheduling issues, the study team was not able to do the psych testing on 2 control participants, this applies to all outcome measures with 142 controls instead of 144.
Measure: Mean (Standard Deviation); unit: number of patterns completed correctly
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
number of patterns completed correctly
  Spatial Span Forward | 9.88 (3.11) | 9.90 (3.22)
  Spatial Span Backward | 10.6 (2.74) | 10.32 (2.84)

4. Primary Outcome: Executive Functioning in Verbal Domain Using A Developmental NEuroPSYchological Assessment-II (NEPSY-II) - Number of Words Generated
Description: The word generation subtest is designed to assess verbal productivity through the ability to generate words within specific semantic and initial letter categories. The participant is given a semantic or initial letter category and asked to produce as many words as possible in 60 seconds. Scores represent the number of words generated and higher scores indicate better executive control of language production, better inhibition and ideation, or better vocabulary knowledge.
Time Frame: Baseline
Population: Only participants aged 7 to 12 were administered this assessment; there is not a version of this test for 6 year olds. Therefore number of subjects analyzed is different from number of enrolled
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 177 | 123
Number of words | 7.21 (2.99) | 7.47 (3.23)

5. Primary Outcome: Planning Ability in the Visual-Spatial Domain Using A Developmental NEuroPSYchological Assessment-II (NEPSY-II): Route-Finding Score
Description: The route finding subtest is designed to assess knowledge of visual spatial relations and directionality, as well as the ability to use this knowledge to transfer a route from a simple schematic map to a more complex one. The participant is shown a schematic map with a target house and asked to find that house in a larger map with other houses and streets. Scores could range from 0 to 20 with higher scores indicating better performance with visuospatial relations and orientation.It's broken into percentile categories: <2% =1, 2-10%= 2, 11-25%=3, 26-75%=4, >75%=5. The scores from the percentile categories described are reported. Higher numbers in the percentile categories indicate better performance with visuospatial relations and orientation.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentile categories
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
percentile categories | 4 [4 to 5] | 4 [4 to 5]

6. Primary Outcome: Behavior Rating Inventory of Executive Function (BRIEF) Score
Description: Behavior Rating Inventory of Executive Function (BRIEF) is a questionnaire composed of three indices: Global Executive Composite, Behavioral Regulation Index, and Metacognition Index. Items are rated in a Likert-scale with 1 (never), 2 (sometimes), and 3 (often). The Global Executive Composite consists of 72 items with scoring ranging from 72 to 216. The Behavioral Regulation Index score is the total of 28 items and ranges from 28 to 84. The Metacognition Index score is the total of 44 items and ranges from 44 to 132. Raw scores are standardized to t-scores with a mean of 50 with a standard deviation of 10. Scores above 50 suggest increased difficulty while scores under 50 reflect better functioning.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
t-score
  Global Executive Composite Index: number analyzed (Participants) | 205 | 142
  Global Executive Composite Index | 51.72 (10.83) | 52.22 (11.54)
  Behavioral Regulation Index | 51.68 (11.56) | 51.49 (11.94)
  Metacognition Index: number analyzed (Participants) | 205 | 142
  Metacognition Index | 51.35 (10.81) | 52.29 (11.44)

7. Primary Outcome: Wechsler Abbreviated Scale of Intelligence-II (WASI-II): Vocabulary Score
Description: The WASI-II: Vocabulary subtest is a quick estimate of an individual's level of intellectual functioning. The subtest is comprised of 42 total items that require the subject to orally define 4 images and 37 words presented both orally and visually. Scores are scaled to a t-score with a mean of 50 and standard deviation of 10. Scores above 50 indicate greater intellectual ability.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
t-score | 56.20 (9.45) | 56.67 (8.57)

8. Primary Outcome: Wechsler Abbreviated Scale of Intelligence-II (WASI-II): Matrix Reasoning Score
Description: The WASI-II: Matrix Reasoning subtest is a quick estimate of an individual's level of intellectual functioning. The subtest is comprised of 35 incomplete grid patterns that require the participant to select the correct response from five possible choices. Scores are scaled to a t-score with a mean of 50 and standard deviation of 10. Scores above 50 indicate greater intellectual ability.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
t-score | 52.44 (9.27) | 52.77 (9.59)

9. Primary Outcome: Brain Wave Latency Assessment Value
Description: The ABER measures the initial response of the auditory pathway to sounds by quantifying the cranial nerve 8 conduction and brain wave latency and amplitude. Three electrodes were attached, one on the forehead and one on each earlobe, to assess response to stimulation. Responses to a clicking sound are recorded by a computerized system.There is not a normative expected range - higher scores mean that the signal is being conducted slower and lower values means that it is being conducted faster.
Time Frame: Baseline
Population: Number of subjects were unable to be scored due to data collection issues(6 cases and 6 controls). Of those that were analyzed, not all of wave latencies were interpretable- which is why the numbers are different. Often wave 1 latency data would not be interpretable, and so would not have a score, but waves 3 and 5 were readable and scored.
Measure: Mean (Standard Deviation); unit: ms (milliseconds)
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 200 | 138
ms (milliseconds)
  Wave 1 Latency: number analyzed (Participants) | 163 | 118
  Wave 1 Latency | 1.69 (0.22) | 1.70 (0.20)
  Wave 3 Latency: number analyzed (Participants) | 194 | 133
  Wave 3 Latency | 3.29 (0.20) | 3.27 (0.20)
  Wave 5 Latency | 5.98 (0.29) | 5.98 (0.31)

10. Primary Outcome: Number of Participants Who Failed Pure-tone Hearing Assessment
Description: Pure-tone hearing test measures both conductive and sensorineural hearing loss. In this procedure, sounds are presented at different frequencies and volumes through speakers, headphones, and small devices placed behind the ear while the participant stands in a soundproof booth. Pass "1" / Fail "2", scores are presented as % of case/control who failed the hearing screen. Hearing was screened in the right and then left ear at 500, 1000, 2000, and 4000 Hz at 30 DB using pure tones in a non-sound proof room. A child received a "1" if s/he responded to all frequencies in both ears and a "2" if s/he did not respond with 2 attempts at one or more frequencies.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
Participants | 12 | 6

11. Primary Outcome: Diagnostic Evaluation of Articulation and Phonology (DEAP) Score
Description: The DEAP evaluates both articulation and phonological processes. The DEAP includes a Diagnostic Screen, a diagnostic Articulation Assessment, a diagnostic Phonology Assessment (with a phonological analysis), and an Oral Motor Screen. The Diagnostic Screen can determine whether a child has a speech difficulty. If all words were produced at least twice (2 of 3 possible trials), there were 25 targets available (25 points possible). Any difference across the 3 trials for 1 word counted as 1 point. For example, 4 instances of words produced differently is 4/25 = 16% occurrence. The test establishes "inconsistent production" at greater than or equal to 40%.
Time Frame: Baseline
Population: There were 7 cases and 16 controls with missing scores-23 total. The reasons were: Missing or Incomplete audio files for scoring reference (21), participant not following instructions (1), and excessive static in background, file inaudible (1).
Measure: Mean (Standard Deviation); unit: percentage of Inconsistent word producti
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 199 | 128
percentage of Inconsistent word producti | 0.06 (0.08) | 0.06 (0.08)

12. Primary Outcome: Diadochokinetic (DDK) Speech Rate
Description: The Diadochokinetic (DDK) speech rate assesses speech and language problems. The DDK rate measures how quickly a participant can say a series of sounds. Scores are second/syllable. Lower value = faster talker. Lowest value of 2-3 trials, or only 1 trial provided/audible.
Time Frame: Baseline
Population: Missing/incomplete audio recording from 5 participants
Measure: Mean (Standard Deviation); unit: second/syllable
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 204 | 141
second/syllable | 0.162 (0.024) | 0.167 (0.024)

13. Primary Outcome: Acoustic Voice Quality Index (AVQI) Score
Description: The Acoustic Voice Quality Index (AVQI) uses multiple acoustic markers to assess dysphonia. Scores can range from 0 to 10 and scores from 0 to 3 suggest normophonia while 10 represents severe dysphonia.
Time Frame: Baseline
Population: Scores for 5 cases and 3 controls were not collected due to excessive ambient noise in the background of the recording interfering with audio quality.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 201 | 141
score on a scale | 3.23 (1.62) | 3.00 (1.78)

14. Primary Outcome: Oral and Written Language (2nd Edition (OWLS-II): Listening Comprehension (LC)) Scales Score
Description: The OWLS-II: LC measures oral language reception, which is the understanding of spoken language. The examiner orally presents increasingly difficult words, phrases, and sentences to the participants and he/she responds by pointing to or stating which of the four pictures is correct. The raw score of the number of correct responses is converted to a standard score based on age. The mean standard score for this test is 100, with a standard deviation of 15 and a range of 50-150, with higher scores indicating better listening comprehension.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale | 102.72 (12.38) | 100.72 (11.85)

15. Primary Outcome: Oral and Written Language (2nd Edition (OWLS-II): Oral Expression (OE)) Scales Score
Description: The OWLS-II: LC measures oral language expression, which is the use of spoken language. The examiner orally presents a verbal prompt along with a picture and the participant must respond orally to the prompt with increasingly difficult language. The raw score of the number of correct responses is converted to a standard score based on age. The mean standard score for this test is 100, with a standard deviation of 15 and a range of 50-150, with higher scores indicating better listening comprehension.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale | 100.85 (13.07) | 98.45 (14.03)

16. Primary Outcome: Movement Assessment Battery for Children-2 (Movement ABC-2): Performance Test Percentiles
Description: Movement ABC-2: Performance test is designed to identify and describe impairments in motor performance of children and adolescents 3-16 years of age. The Performance Test involves children completing a series of fine and gross motor tasks grouped into three categories: Manual Dexterity, Aiming and Catching, and Balance. A tester will observe and record how the child performs the task. The scores are given in percentiles, with 50% being the average score- below 50% means below average, and a range of 1%-99%. Children whose performance falls below the 15th percentile may benefit from intervention, with those between the 6th and 15th percentile being at risk for Developmental Coordination Disorder (DCD). Those whose performance is at or below the 5th percentile represent children with DCD if other criteria are also met.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
Percentile | 43 (30) | 43 (31)

17. Primary Outcome: Iowa Oral Performance Instrument (IOPI) Tongue Strength Value
Description: IOPI is a hand held manometer which measures intraoral pressure generated by compression of an air filled bulb by the tongue against the palate. Strength is measured in kilopascal (kPa). Typically, tongue strength is decreased in subjects with classic galactosemia and can contribute to speech disorders.
Time Frame: Baseline
Population: There are fewer participants for this outcome measure - these children have dental/orthodontic fixed wires over the roof of their mouth that made it impossible to do this task.
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 202 | 139
kilopascal (kPa) | 55.41 (13.14) | 55.02 (12.63)

18. Primary Outcome: Essential Tremor Rating Assessment Scale (TETRAS) Score
Description: TETRAS consists of 10 items that evaluate tremor in the head, arms, and legs. The rater assigns a score of 0 to 4 for each item, in ascending order of severity. Total scores range from 0 to 40 with higher scores indicating greater severity of tremors.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale | 26.41 (7.06) | 26.46 (7.19)

19. Primary Outcome: Social Skills Improvement System (SSIS) Rating Scales Score
Description: The SSIS is a parent-reported measure that evaluates Social Skills and Problem Behaviors. 38 items are rated in a Likert-scale of 0 (never) to 3 (very often). The raw scores are converted to scaled scores with a mean of 100, a standard deviation of 15, and a range of 50-150. Standard scores are derived from the scores of a large nationally representative sample of individuals having a similar age and the same sex. Higher standard scores for "Social Skills" indicate more positive social skills, while higher standard scores for "Problem Behaviors" indicates more maladaptive behaviors (i.e. lower scores indicate fewer problem behaviors).
Time Frame: Baseline
Population: This was a parent survey. Four were unable to be scored because they were incomplete (2 cases and 2 controls) and 1 case survey that had the social skills section complete but the problem behaviors section incomplete, so could only be partially scored.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 204 | 142
score on a scale
  Social Skills Standard Score | 97.68 (13.45) | 98.08 (14.07)
  Problem Behaviors Standard Score: number analyzed (Participants) | 203 | 142
  Problem Behaviors Standard Score | 98.85 (49.06) | 98.12 (13.99)

20. Primary Outcome: Child Behavior Checklist for Ages 6-18 (CBCL/6-18) T-Scores
Description: The CBCL is a parent-reported measure that evaluates a child internalizing and externalizing behaviors and total problems. It consists of 140 questions on a Likert-scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. Total raw scores are converted to t-scores with a mean of 50 and standard deviation of 10. Higher scores indicative of better behavior and less problems.
Time Frame: Baseline
Population: These were parent surveys and 4 surveys were not completed (forgot back page) and they did not respond to requests later to complete it.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 202 | 144
t-score | 49.06 (11.02) | 49.40 (11.44)

21. Primary Outcome: Revised Children's Manifest Anxiety Scale-2nd Edition (RCMAS-2) T-Scores
Description: RCMAS measures for the presence of academic stress, test anxiety, peer and family conflicts, and drug problems in children. The test consists of 49 yes/no items and a total score is calculated by summing the number of yes responses. The total raw score is converted to a t-scores with a mean of 50 and a standard deviation of 10. Scores above 60 generally indicate that the child is experiencing some level of anxiety.
Time Frame: Baseline
Population: Unable to collect this measure on one child due to scheduling restraints
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 143
t-score | 46.27 (9.98) | 46.66 (11.14)

22. Primary Outcome: Number of Children Participating in Special Education or Other Intervention Experiences
Description: Questionnaire developed by project staff based on experiences of children, as reported by parents, with classic galactosemia with questions on specific problems experienced, when identified, placement or intervention, other problems.
Time Frame: Baseline
Population: These questions were part of a survey administered to parents prior to part 2 testing, 4 of these surveys gave incomplete answers to these questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 204 | 143
Participants | 44 | 30

23. Primary Outcome: Pediatric Adventitious Movement Scale - Upper Extremity Steadiness Score
Description: The upper extremity steadiness assessment is the "dot task", where subjects are asked to hover a pen/stylus a dot steadily for 20 seconds without touching the page/screen and keeping the arm/elbow lifted off the table. Movement in the X, Y, and Z dimensions (left-right, up-down, vertical movement) are recorded on video and scored by overlaying a measurement onto the video to determine the extent of adventitious movement. A lower score indicates increased upper extremity steadiness, with 0 being no movement.
  0 = no adventitious movement,
  1. = adventitious movement is barely visible, 1.5 = adventitious movement is visible, but less than 1 cm,
  2. = adventitious movement is 1- < 3 cm amplitude, 2.5 = adventitious movement is 3- < 5 cm amplitude,
  3. = adventitious movement is 5- < 10 cm amplitude, 3.5 = adventitious movement is 10- < 20 cm amplitude,
  4. = adventitious movement is > 20 cm amplitude.
Time Frame: Baseline
Population: There were 2 children who had prior broken arms/injuries to the left hand that could only do the test on the right hand side.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale
  Right hand | 1.5 (0.52) | 1.45 (0.52)
  Left hand: number analyzed (Participants) | 205 | 143
  Left hand | 1.67 (0.56) | 1.64 (0.56)

24. Primary Outcome: Pediatric Adventitious Movement Scale - Archimedes Spiral Task Measurement
Description: This measure involves using a stylus pen to draw an Archimedes spiral in between the lines of a spiral template that is displayed on the tablet screen. The drawn spiral is recorded by the Neuroglyphics software on a SurfacePro3 tablet which displays the spiral template and records position and pressure of the pen tip as the subject draws. The pen should be held such that no part of the hand or arm touches the table. The scoring for this measure is the root mean square (RMS) of the drawn spiral compared to the "ideal" spiral. The root mean square is the square root of the arithmetic mean of the squares of a set of numbers representing the distance between processive points on an actual spiral drawn by a participant and what would have been an "ideal spiral" drawn mid-way between the template outlines provided on the tablet. The closer the drawn spiral was to the "ideal spiral" the smaller the RMS value will be.
Time Frame: Baseline
Population: The study team had significant technical issues with this program and so it did not work at all for a number of testing blocks, resulting in a much smaller number of participants collected.
Measure: Mean (Standard Deviation); unit: root mean square (in millimeters)
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 165 | 109
root mean square (in millimeters)
  Right hand | 130.55 (61.90) | 132.41 (68.69)
  Left hand | 145.37 (56.78) | 145.48 (68.22)

25. Primary Outcome: Hand Strength Value
Description: Hand strength will be assessed with a standard pediatric dynamometer. Pediatric reference ranges for hand strength vary depending on age and gender; for this study the hand strength of cases and controls are compared.
Time Frame: Baseline
Population: One control was not able to be collected due to a broken hand/arm in a cast (could not complete task).
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 143
kilograms | 15.49 (5.03) | 15.55 (4.69)

26. Primary Outcome: The Goldman Fristoe Test of Articulation-3 (GFTA-3) Score
Description: The Goldman Fristoe Test of Articulation-3 (GFTA-3) is a systemic measure of articulate consonant and vowel sounds for children. The average standard score for this test is 100, with a standard deviation of 15 and a range of 50-150, with higher scores indicating better articulation. The raw score of the number of speech errors during the test, and is converted to a standard score based on age and sex.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale | 88.95 (21.91) | 88.79 (22.77)

27. Primary Outcome: The Children's Depression Inventory-2 (CDI-2) Score
Description: The Children's Depression Inventory-2 (CDI-2) is a screening measure for symptoms of depression in children. It is a self-report form and includes 12 items. Each item receives a score of 0-2, where 0 = the absence of depressive symptoms and 2 = definite symptoms of depression. Total raw scores are converted to t-scores, with a mean of 50 and a standard deviation of 10. T-scores between 45 and 55 are generally considered normal and higher scores indicates more depressive symptoms.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 142
t-score | 53.82 (12.04) | 53.08 (11.35)

28. Primary Outcome: Structure-Function-Praxis (SFP) Exam Score
Description: SFP is a non-standardized 53-item exam of the oral and facial structures (Structure), the range and speed of movement of the oral and facial structures (Function), and the ability to imitate non-speech single and sequential movements (Praxis). The Structure score had a range of 0-10, with 10 items scored as "0"-within functional limits, or "1"-deviant. The Function score had a range of 0-66, consisting of 33 items scored as "0"- within functional limits, "1"- mild/moderate impairment, or "2"- severe impairment. The Praxis score had a scale from 0-40, and consisted of 10 items scored as "0"- imitates immediately, "1"- mild groping; or delayed but successful, "2"- groping or sequential efforts, then success, "3"- could not achieve imitation with purposeful effort, or "4"- child does not/cannot attempt the task. The scores from the three domains are summed to create an overall SFP score, with a possible range of 0 -116. For this exam, the closer to zero, the better the score.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
Number analyzed (Participants) | 206 | 144
score on a scale | 8.09 [0 to 25] | 8.13 [0 to 37]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the direct testing visit (Day 1). Due to the nature of this observational study, no adverse events were anticipated.
Description: Adverse event reporting includes all participants who attended the direct testing visit, regardless of if complete information was collected during this visit.
Arm/Group | Children With Duarte Galactosemia (Cases) | Unaffected Siblings (Controls)
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/149
Other Adverse Events (participants affected / at risk) | 0/212 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02519504/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT02519504/SAP_001.pdf